CLINICAL TRIAL: NCT00147862
Title: Does Tranexamic Acid Administration Reduce Blood Loss During Head and Neck Surgery?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMH/185/IM-2004; TMH/185/IM-2004
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Head and Neck Neoplasms
Keywords: Tranexamic Acid; Antifibrinolytic Agents; Head and Neck Neoplasms; Thromboelastography
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid

SUMMARY:
To Study whether infusion of Tranexamic Acid (a synthetic antifibrinolytic agent) reduces blood loss during head and neck surgery.

DETAILED DESCRIPTION:
Blood and blood products are precious resources. Administration of blood and blood product carries with it the risk of postoperative bacterial infection1 and increased recurrence rates in certain types of cancers. Lower transfusion trigger, preoperative autologous blood donation with or without erythropoietin, intraoperative red blood cell salvage, regional anesthesia, controlled hypotension, and antifibrinolytic agents are all useful means to decrease the need for allogenic transfusions.

Tranexamic acid, a synthetic antifibrinolytic agent that binds to the lysine binding site of plasminogen and blocks the binding of plasminogen to the fibrin surface. Thus plasminogen activation is prevented and fibrinolysis is delayed. It has been used to reduce blood loss during coronary revascularization, orthotopic liver transplantation4, scoliosis correction surgery and other orthopedic procedures. The use of tranexamic acid intraoperatively has been shown to reduce blood loss by 25 - 40% in various studies. The primary concern when administering an antifibrinolytic drug is the potential increased incidence of thromboembolic events. A common misconception is that synthetic antifibrinolytic drugs increase blood clotting. The drugs do not alter blood clotting, but rather slow dissolution of blood clots. There is no data on the utility of tranexamic acid to reduce blood loss in head & neck cancer surgery.

We wanted to compare Tranexamic Acid infusion to Saline (Placebo)infusion to see whether Tranexamic ACid Administration will reduce blood loss. Reduction in transfusion requirements will lead to reduced costs and possible reduction in complications of blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* All eligible previously untreated patients with resectable squamous cell carcinoma of the oral cavity
* Undergoing composite resection of the mandible along with neck dissection and requiring reconstructive procedures in the form of pedicled flaps.
* Patients who agree to participate by giving informed consent.

Exclusion Criteria:

* Coagulopathy form any cause (Abnormal coagulogram - prothrombin time (PT) > 18 seconds or partial prothrombin time (PTT) > 50 seconds, recent (<5 days) acetylsalicylic acid ingestion, anticoagulant therapy (heparin, 4 hours preoperative or warfarin, 3 days preoperatively).
* Pre-existing renal dysfunction (serum creatinine 200 mmol/L),
* Known allergy to tranexamic acid,
* Peripheral vascular disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2005-05; Study Completion 2007-01

PRIMARY OUTCOMES:
Administration of tranexamic acid reduces perioperative blood loss and thus,
Requirement for replacement of blood in head and neck surgeries

SECONDARY OUTCOMES:
To observe procoagulant effects leading to complications, if any.
Cost effectiveness of the drug in terms of savings on blood transfusion requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Atul P Kulkarni, MD, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India